CLINICAL TRIAL: NCT00448149
Title: Phase I/II Trial of RAD001 Plus Nexavar® For Patients With Metastatic Renal Cell Carcinoma
Brief Title: Phase I/II Trial of RAD001 Plus Nexavar in Patients With Kidney Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PAC IRB#1006-0152; RCC-06-102 (Other: Principal Investigator)
Record Dates: First submitted 2007-03-15; First posted 2007-03-16 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Carcinoma, Renal Cell
Keywords: Kidney cancer; Renal cell carcinoma; Metastatic RCC
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — Everolimus; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): To establish the maximally tolerated dose (MTD) of RAD001 in combination with Nexavar®
  Interventions: Drug: RAD001; Drug: Sorafenib

INTERVENTIONS:
Drug: RAD001 — RAD001 will be administered orally once a day, daily, without interruption per 4 wk cycle for 2 cycles. MTD is established in Phase I portion of trial (2.5, 5 or 10mg). If responding, additional therapy will be given.
  Other Names: Everolimus
Drug: Sorafenib — A dose of 400mg of Nexavar® will be administered orally twice a day, daily, without an interruption per 4 week cycle for 2 cycles. If responding, additional therapy will be given.
  Other Names: Nexavar®, BAY-4900

SUMMARY:
The purpose of this study is to see whether the combination for RAD001 and Nexavar® works better when given together than they do alone. The purpose of the first phase of this study is to determine the best dose of RAD001 given with Nexavar®, and to see what effects, good and/or bad, the study drug has on the subject and the subject's tumor. This study will also observe side effects experienced by the subject.

DETAILED DESCRIPTION:
Despite significant progress in understanding the biology of renal cell carcinoma (RCC), it is estimated that over 35, 000 people in the United States will be diagnosed and approximately 12, 000 have died from this disease in 2005. Renal cell carcinoma presently ranks tenth as the leading cause of cancer death and constitutes 3% of all solid neoplasms.

In contrast to many other malignancies, treatment for RCC is limited. Treatment remains a highly difficult and perplexing challenge due to its resistance to both chemotherapy and hormone therapy and limited response to cytokines. Despite recent advances in our fundamental knowledge of RCC biology and development of molecular therapeutics, more clinical research will be required to best guide our use of these exciting new agents in combination regimens.

The combination of RAD001 and Nexavar®, in current clinical trials with minimal toxicity, represents a treatment regimen which should be investigated for tolerance and toxicity as well as initial phase II efficacy. The study is designed to evaluate the MTD. Following the completion of the phase I, utilizing the MTD, Phase II study is designed to evaluate the anti-tumor activity.

ELIGIBILITY:
Inclusion Criteria:

* Histologic confirmed predominant clear cell renal cell carcinoma.
* Patients must have progressive metastatic disease.
* Paraffin RCC tissue blocks or unstained slides must be available.
* Karnofsky performance status > 70% .
* Not pregnant
* Age > 18
* Initial laboratory values must meet requirements
* Phase I: No more than three prior systemic and/or investigative therapy for MRCC. Previous therapy may include prior single agent exposure to RAD001 or Nexavar®. Four weeks must have elapsed from previous therapy.
* Phase II: No more than one prior systemic and/or investigative therapy of any kind for MRCC. Four weeks must have elapsed from previous therapy.
* Phase II: Previous therapy may not include RAD001 or Nexavar®.
* Phase II: Patients with primary tumor in place are strongly encouraged to undergo nephrectomy prior to initiation of study agent.
* Phase II: Prior palliative radiotherapy to metastatic lesion(s) is permitted. Patient must have adequately recovered from the acute toxicities of this treatment.
* Phase II: All major surgery of any type and/or radiotherapy must be completed at least 4 weeks prior to registration.

Exclusion Criteria:

* No ongoing hemoptysis or cerebrovascular accident within 12 months, or peripheral vascular disease with claudication on less than 1 block, or history of clinically significant bleeding.
* No deep venous thrombosis or pulmonary embolus within one year and no ongoing need for full-dose oral or parenteral anticoagulation.
* No evidence of current central nervous system (CNS) metastases.
* No significant cardiovascular disease
* No patients with uncontrolled hypertension
* Any ongoing requirement for systemic corticosteroid therapy (except replacement therapy for adrenal insufficiency) or other immunosuppressants are not permitted.
* Patients with a pre-existing thyroid abnormality whose thyroid function cannot be maintained in the normal range by medication are ineligible.
* No uncontrolled psychiatric disorder.
* Patients with delayed healing of wounds, ulcers, and/or bone fractures are not eligible.
* Patients with a 'currently active' second malignancy other than non-melanoma skin cancers are not eligible. Patients are not considered to have a 'currently active' malignancy if they have completed anti-cancer therapy and are considered by their physician to be a less than 30% risk of relapse.
* Pregnant women are excluded
* All fertile patients must use adequate contraception (barrier method) while on study and for three months thereafter. Oral, implantable, or injectable contraceptives may be affected by cytochrome P450 interactions, and are therefore not considered effective for this study.
* Prior treatment with any investigational drug within the preceding 4 weeks.
* Other concurrent severe and/or uncontrolled medical disease which could compromise participation in the study (i.e., uncontrolled diabetes, severe infection, severe malnutrition, ventricular arrhythmias, chronic liver or renal disease, active upper GI tract ulceration).
* A known history of HIV seropositivity.
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of RAD001 (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2006-12; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Phase I: To establish the maximally tolerated dose (MTD) and safety profile of RAD001 in combination with Nexavar® in patients with metastatic renal cell carcinoma (MRCC). | 1 year
Phase II: Study the anti-tumor effects of RAD001 plus Nexavar® | 2 years

SECONDARY OUTCOMES:
Phase II: Response rate | restaging every 8 weeks
Duration of tumor response | restaging every 8 weeks
Progression free survival | restaging every 8 weeks
Overall survival | restaging every 8 weeks
Study the safety of RAD001 plus Nexavar® given at MTD. | AEs as occur

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Amato, DO, Principal Investigator — Baylor College of Medicine - Methodist Hospital
Locations (1):
- The Methodist Hospital Research Institute, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No